CLINICAL TRIAL: NCT06438406
Title: Postural Assessment, Therapeutic Exercise and Orthotic Devices in the Prevention of Haemophilic Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MFR052024
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Haemophilic Arthropathy; Orthosis; Foot Malalignment
Keywords: haemophilic arthropathy; orthosis; postural assestment; foot malalignment; therapeutic exercise; haemarthroses; haematomas; HJHS; FISH
MeSH Terms: conditions — Hematoma | interventions — Orthotic Devices; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthotic devices and therapeutic exercise (Group A) (Active Comparator): Group A consisting of patients who were prescribed orthoses, to use gradually, and a 20-session rehabilitation programme, based on the Back School method
  Interventions: Device: Orthotic devices and therapeutic exercise (Group A); Device: Orthotic devices (Group B)
- Orthotic devices (Group B) (Active Comparator): Group B consisting of patients who were only prescribed orthoses for the lower limbs
  Interventions: Device: Orthotic devices and therapeutic exercise (Group A); Device: Orthotic devices (Group B)

INTERVENTIONS:
Device: Orthotic devices and therapeutic exercise (Group A) — Group A consisting of patients who were prescribed orthoses, to use gradually, and a 20-session rehabilitation programme, based on the Back School method
Device: Orthotic devices (Group B) — Group B consisting of patients who were only prescribed orthoses for the lower limbs

SUMMARY:
Haemophilic arthropathy (HA) is the most frequent complication of haemophilia and is often associated with a severe deterioration in quality of life. It is caused by repeated joint bleeding resulting in chronic proliferative synovitis and progressive destruction of articular cartilage. The most frequently affected joints are the knees, ankles and elbows.

The aim of this study is to verify the use of lower limb orthoses in combination with postural rehabilitation, assessing the incidence of spontaneous haemarthroses and haematomas as the primary endpoint and pain and QoL as secondary endpoints.

We conducted a prospective observational, randomised and controlled study on outpatients attending the UOC of Recovery and Functional Rehabilitation of the AOUP Paolo Giaccone of Palermo for haemophilic arthropathy sent by the UO of Haematology of the same hospital. The study period was between January 2017 and March 2023.

The patients recruited were randomly divided into two groups by means of a computer-generated random number system: group A, consisting of patients who were prescribed orthoses and a 20-session rehabilitation programme; group B, consisting of patients who were only prescribed orthoses for the lower limbs. The rehabilitation programme was based on the Back School method.

All patients were assessed at baseline (T0), at 3 months (T1) and after 6 months (T2).

Two arthropathic-specific scales were used to assess outcomes, namely the Hemophilia Joint Health Score (HJHS), which reflects joint function and status, and the Functional Independence Score in Hemophilia (FISH), which relates to the patient's quality of life. We also used the Numerical Rating Scale (NRS) for joint pain. Finally, postural assessment was performed in static posture, observing the patient's alignment in different planes and using the APECS (AI Posture Evaluation and Correction System ®) mobile app. During the re-evaluations, any new haemarthroses and haematomas were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe haemophilia A or B;
* age ≥ 6 years and ≤ 50 years;
* presence of hindfoot and/or arch misalignment;
* prophylaxis with factor deficient (VIII or IX).

Exclusion Criteria:

* patients with prosthetic implants/synthetic means
* uncooperative patients

Ages: 6 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
prevention of haemophilic arthropathy | All patients were assessed at 3 months (T1) and after 6 months (T2).
  During re-evaluations, the possible appearance of new haemarthroses and haematomas was assessed ,which were absent at the baseline examination

SECONDARY OUTCOMES:
Functional Independence Score in Hemophilia (FISH) | All patients were assessed at baseline (T0), at 3 months (T1) and after 6 months (T2)
  This score is a performance-based assessment tool used to measure the functional ability of patients. The maximum score is 32 (the greatest autonomy).
Hemophilia Joint Health Score (HJHS) | All patients were assessed at baseline (T0), at 3 months (T1) and after 6 months (T2)
  The Hemophilia Joint Health Score is a rating scale that measures joint health in the domains of anatomical structure and function (biomechanics) of the joints most frequently affected by haemorrhage in haemophilia: knees, ankles, elbows.
Numerical Rating Scale (NRS) | All patients were assessed at baseline (T0), at 3 months (T1) and after 6 months (T2)
  The NRS scale is a one-dimensional 11-point scale that assesses pain intensity in adults, with a range from 0 to 10, corresponding to 'no pain' and 'worst pain imaginable'

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: https://www.unipa.it/persone/docenti/l/giulia.letiziamauro/